CLINICAL TRIAL: NCT01180283
Title: Efficacy and Safety of Lodenafil Carbonate in the Treatment of Erectile Dysfunction in Patient With Type II Diabetes. Multicentric Study.
Brief Title: Efficacy and Safety of Lodenafil Carbonate in the Treatment of Erectile Dysfunction in Patients With Diabetes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Jorge Barros Afiune, CRISTÁLIA PRODUTOS QUÍMICOS FARMACÊUTICOS LTDA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRIST 002
Record Dates: First submitted 2010-07-29; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Lodenafil carbonate; Diabetes
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus | interventions — lodenafil carbonate

ARMS (1):
- lodenafil carbonate (Helleva®) (Experimental)
  Interventions: Drug: lodenafil carbonate

INTERVENTIONS:
Drug: lodenafil carbonate — Dosage: lodenafil carbonate 80mg once a day. It should be taken between 6 and 2 hours before the sexual intercounter.

SUMMARY:
Sixty diabetes men with erectile dysfunction from mild to severe who agree to participate is going to have medical care approximately for 16 weeks.

During the first 4 weeks, patients will not receive any inhibitor of phosphodiesterase 5. In the following eight weeks, patients will receive oral lodenafil carbonate. They will complete the International Index of Erectile Dysfunction (IIEF) questionnaire in the site and answer the Sexual Encounter Profile (SEP) questions 2 and 3 and the Erection Hadness Score (EHS) after each intercourse or attempt without or using oral lodenafil cardonate 80mg.

Questionnaire of adverse event is included in patient diary.

DETAILED DESCRIPTION:
This is a prospective, fixed dose, open label study.

The run in period from inclusion to conclusion will be between fourteen and sixteen weeks.

Visit zero (Vo):

* Patients will sign the informed consent form;
* Investigator will clinically evaluate the subjects regarding eligibility criteria;
* Safety laboratory tests will be perform ;
* Patients will answer the erectile function domain of the International Index of Erectile Function (IIEF);

Study coordinator:

Will orientate subjects regarding the follow:

* Patients will not use any phosphodiesterase- 5 inhibitor (iPDE-5) for four weeks;
* When intercourse or attempt happen, subjects will fill a diary;

Patients' diary includes: questions 2 and 3 of Sexual Encounter Profile (SEP), the Erectile Hardness Score (EHS) and adverse events data.

Subject will return after four weeks.

Visit One (V1):

* Patients will answer basal IIEF;
* Investigator will inform to patient the laboratory tests results;

Study coordinator:

* Will give to the patients eight pills of lodenafil carbonate;
* Will give instructions about study medication; Patient should take one pill from six to two hours before intercourse or attempt, with or without food intake or drink. The patient will not take more than one pill daily.
* When intercourse or attempt happen, subjects will fill out the diary; Patients' diary includes: questions 2 and 3 of Sexual Encounter Profile (SEP), the Erectile Hardness Score (EHS) and adverse events data.

Subject will return after four weeks.

Visit two (V2)

Study coordinator:

* Will give to patient eight pills of lodenafil carbonate;
* Will give instructions about study medication:

Patient will take one pill from six to two hours before intercourse or attempt, with or without food intake or drink. The patient will not take more than one pill daily.

- When intercourse or attempt happen, subjects will fill out the diary;

Patients' diary includes: questions 2 and 3 of Sexual Encounter Profile (SEP), the Erectile Hardness Score (EHS) and adverse events data.

Subject will return after four weeks.

Visit three (V3)

* Patients will answer the International Index of Erectile Function (IIEF);
* Safety laboratory will be perform ;

Visit four (V4)

- Investigator will inform to patients the laboratory tests results;

Complete medical evaluation including adverse event questions and physical examinations will be done at all visits.

Efficacy will be assessed by files of patients who complete the study and did not have protocol violation (per protocol population).

Main outcomes to measure efficacy: IIEF (questions 1 to 15), SEP question 2 (Were you able to insert your penis into your partner's vagina?), SEP question 3 (Did your erection last long enough for you to have successful intercourse?), EHS (Erection Hardness Score).

Tolerability will be assessed by files of patients intend to treat - subjects who took the study medication at least once.

Patients logs contain questions such as: Did you experience any uncomfortable symptoms?; At what time this symptoms began?; Did you take medication to relieve the symptoms?; Did you go to the hospital /or doctor's office?.

After review the logs, investigator will interview patients to fill adverse events reports. Investigator will assess the event intensity (from mild to severe) and will define the casual relationship to the study medication (definite; probable; possible; doubtful).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type II;
* Age from 18 to 65 years;
* Erectile dysfunction within the previous 6 months;
* Mild, moderate or severe erectile dysfunction by IIEF questionnaire;
* Stable sexual partner in the past 2 months;
* Preserved libido;
* Studied at least up to fourth grade;

Exclusion Criteria:

* Current beta blocker, thiazide, alpha methyldopa, antidepressants, or antiandrogen therapy intake;
* Penile prosthesis;
* Previous intolerance to sildenafil, vardenafil, tadalafil or lodenafil carbonate;
* Previous negative response to iPDE-5 correct use.;
* Penile anatomical deformities;
* Previous penile surgeries for erectile dysfunction, premature ejaculation or penile enlargement;
* Myocardial infarction or cerebral vascular accident within the previous 6 months;
* Severe or uncontrolled cardiac diseases;
* Spinal cord injury, multiple sclerosis, retinitis pigmentosa;
* Radical pelvic surgery and pelvic radiotherapy, including radical prostatectomy;
* Myocardial or Coronary Artery disease with cardiologist contraindication for using iPDE5;
* Cancer;
* Anaphylactic reactions or Steven-Johnson disease;
* Participation in another clinical trial within the last 2 months;
* Sexually transmitted diseases;
* Glycated hemoglobin > 12%;
* Testosterone < 200ng/dL;
* Prolactin > 20ng/dL;
* Hemoglobin < 10g/dL;
* Leucocytes > 14.000 cel/mm3;
* TGO > 100 U/L;
* TGP > 100 U/L;
* Creatina > 2 mg/dL;
* Investigator´s opinion;

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-01; Study Completion 2010-04

PRIMARY OUTCOMES:
Evidence that lodenafil carbonate improves erectile function in patients with diabetes type 2. | 16 mounths
  Efficacy is assessing by files of patients including questionnaires like IIEF, SEP and EHS.

SECONDARY OUTCOMES:
Adverse events in type 2 diabetes patients taking lodenafil carbonate and laboratory tests changes after this treatment. | 16 months
  Investigator will interview patients to fill adverse events reports.
  Laboratory tests results before and after lodenafil carbonate treatment will be analyzed and compared, in order to detect significant changes.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital do Servidor Público Estadual de São Paulo, São Paulo, São Paulo
  - Hospital Ipiranga, São Paulo, São Paulo